CLINICAL TRIAL: NCT04954261
Title: Implementing Delirium Detection in Pediatric Intensive Care Unit Through a French Translation of the CAPD : a French Monocentric Observational Study
Brief Title: Delirium Detection in Pediatric Intensive Care Unit Through a French Translation of the CAPD : a French Monocentric Observational Study
Acronym: DeliReP
Status: Withdrawn | Type: Observational
Why Stopped: Abandoned study project
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI18018J; 2018-A00763-52 (Other: ID-RCB)
Record Dates: First submitted 2018-09-07; First posted 2021-07-08 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2021-12

CONDITIONS: Delirium
Keywords: Delirium; paediatric intensive care unit; CAPD (Cornell Assessment of Paediatric Delirium); French translation
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: CAPD — CAPD evaluation every day per 12hours during their stay in PICU

SUMMARY:
The purpose of this study is to introduce delirium detection and try to determine the prevalence of delirium in Pediatric Intensive Care Unit (PICU) using a validated tool : the Cornell Assessment of Pediatric Delirium (CAPD) for every patient twice a day.

DETAILED DESCRIPTION:
Delirium is a frequent affection in ICU. In adult population, its prevalence is 20-50% in non intubated patients and 60-80% in patients under invasive ventilation. It is also frequent in paediatric population, but less diagnosed, whereas it can lead to higher duration stay, higher morbidity, traumatic injuries, acute stress, memory losses and post-traumatic stress syndrome. Since 2016, international guidelines recommend to look for delirium in paediatric population in PICU. There are 3 recommended tools to diagnose this affection: psCAM-ICU (6 months-5 years old), pCAM-ICU (5 years old-18 years old) and CAPD (birth-18 years old).

None of these validated tools have been translated in French.

The principal objective is to study the practicability of twice a day detection of delirium in PICU using the CAPD.

Investigators will first used a validation process to translate the CAPD in French, based on the validation method for psychological questionnaires suggested by Vallerand.

Then they will ask the paramedics to evaluate through the CAPD every consecutive patient/12 hours, every day during their stay in PICU, except for those completely unresponsive or under curare. This systematic evaluation will take place for 2 consecutive months.

For every patient, data will be collected about their age, sexe, term of birth, mental affection status, diagnosis at entry, and daily risk of mortality score, length of stay, ventilation, pain evaluation and treatment, withdrawal evaluation, surroundings, use of hypnotic treatment, steroids, opioids and ketamine.

The secondary aims are to determine the prevalence of delirium with the data collected, to ask whether or not the French version of CAPD has been easily and correctly used, can help to diagnose delirium, and whether investigators can find some associated parameters to delirium.

ELIGIBILITY:
Inclusion Criteria:

* Being hospitalized in PICU during the inclusion period
* Age 0 to 18 years old

Exclusion Criteria:

* Patient with a state of sedation that does not allow the assessment of a change in the state of consciousness or cognitive functioning (equivalent score Richmond Agitation-Sedation Scale RASS <-3 or COMFORT B <11)
* Patient or Parental opposition to the observational study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients aged 0 to 18 years hospitalized in PICU at Necker Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2018-12-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of delirium in the PICU population | 2 months
  Number of CAPD evaluated > 9 / total number of CAPD evaluated

SECONDARY OUTCOMES:
Applicability of the CAPD by the paramedics | Before inclusion period
  5 questions :
  1. Whether or not they have already heard about delirium
  2. Whether or not they know the symptoms of delirium in children and adolescents
  3. Whether or not they have already been confronted to a state of delirium in the Pediatric Intensive Care Unit
  4. Whether of not they think it would be useful to have a specific scale to diagnose delirium in the Pediatric Intensive Care Unit
  5. Whether or not they think it would be feasible to use such a scale regularly in the Pediatric Intensive Care Unit The proposed answers will be Yes, No or I don't know for each question The analysis will be qualitative and quantitative.
Applicability of the CAPD by the paramedics after the 2 months period | 2 months
  The same 5 questions of the pre-test, 5 new closed-ended questions and 3 open-ended questions :
  1. Whether or not they had difficulties evaluating patients with the CAPD
  2. How they evaluate the duration of the evaluation by the CAPD
  3. Whether or not they evaluated the patients with a colleague
  4. Whether or not they think that the assessment of delirium by the CAPD is relevant among PICU patients
  5. Whether or not they think that a long-term evaluation of delirium by the CAPD is feasible in this PICU unit
  1- If difficulties of evaluating patients with the CAPD : quote the difficulties 2- In which categories of patients do they think that the CAPD in not adapted 3- Comment or suggestions to improve the use of the scale
Use of the CAPD by the paramedics | 2 months
  % of CAPD completed during the 2 months period
Age | 2 months
  Potential associated factors to delirium
Sex | 2 months
  Potential associated factors to delirium
Term of birth | 2 months
  Potential associated factors to delirium
Prior neurological impairment | 2 months
  Potential associated factors to delirium
Diagnosis (motivating hospitalization in intensive care) | 2 months
  Potential associated factors to delirium
Severity score on arrival (PIM 3) | 2 months
  Potential associated factors to delirium. Pediatric Index of Mortality (PIM) 3 is a published and open acces program whith 10 variables about the patients (7 binary variables and 3 quantitative ones), that predicts the death probability of the patient. One evaluation per patient at the admission in the PICU unit.
Daily severity score (PELOD 2) | 2 months
  Potential associated factors to delirium. PELOD 2 (PEdiatric Logistic Organ Dysfunction) is a published and open acces program that includes ten variables corresponding to five organ dysfunctions. It predicts a daily percentage of mortality. One evaluation per day per patient during the PICU unit stay.
Duration of hospitalization | 2 months
  Potential associated factors to delirium
Death or survival of the patient | 2 months
  Potential associated factors to delirium
Mechanical ventilation, non invasive ventilation or spontaneous ventilation | 2 months
  Potential associated factors to delirium
Mechanical ventilation time | 2 months
  Potential associated factors to delirium
Presence of parents | 2 months
  Potential associated factors to delirium
Presence of pain | 2 months
  Potential associated factors to delirium.
  Pain was evaluated through the appropriate scale amongst :
  * Comfort B (pediatric behavioural scale, ventilated, sedated and/or comatose patient): seven items scored 1 to 5, a total score greater than or equal to 17/35 indicating a state of pain,
  * or EVENDOL (behavioural scale for conscious patients between birth and 6 years old): five items scored 0 to 3, a total score greater than or equal to 3/15 indicating a state of pain,
  * or FLACC (Face Leg Activity Cry Consolability) (pediatric behavioural scale, usable in patients with cognitive impairment): five items scored 0 to 2, a total score greater than or equal to 3/10 indicating a state of pain,
  Patients able to assess pain felt :
  * Numerical Scale (for patients over 10 years old) a score greater than or equal to 3/10 indicating a state of pain,
  * or Visual Analogue Scale (for patients between 6 and 10 years old), a score greater than or equal to 3/10 indicating a state of pain.
withdrawal or not | 2 months
  Potential associated factors to delirium. Withdrawal was evaluated through the scale WAT-1 (Wthdrawal Assessing tool version 1): ten items scored 0 or 1, and 1 item scored 0 to 2, a total score greater than or equal to 3/12 indicating a state of withdrawal.
Use of benzodiazepines, ketamine, corticosteroids or opioids | 2 months
  Potential associated factors to delirium

CONTACTS AND LOCATIONS:
Overall Officials: Laure De Saint Blanquat, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Necker Enfants Malades Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided